CLINICAL TRIAL: NCT05505721
Title: Do Children and Adolescents With Type 1 Diabetes Have Healthy Eating?:Real-life Data
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Yasemin Atik Altinok, principal investigator, Ege University
Other Study IDs: food diary T1D
Record Dates: First submitted 2022-06-17; First posted 2022-08-18 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Type 1 Diabetes; Children; Adolescent
Keywords: type 1 diabetes; children; adolescents; diet
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to examine the relationship between the nutritional content of the diet consumed by children and adolescents (0-18 years old) with the diagnosis of type 1 diabetes and metabolic control. In this cross-sectional study, 150 children and adolescents with type 1 diabetes who came to Ege University Child Health and Diseases Department, Pediatric Endocrine and Diabetes Department for regular check-ups (4 diabetes control/year) and kept food consumption records in the last 1 year will be included. Body weight and height measurements of the cases will be done by the same person in Ege University Pediatric Endocrinology and Diabetes BD Polyclinic. Turkish Standard Institute approved Baster brand weighing instrument with 0.1 kg intervals and height measurements will be made with Harpander brand stadiometer with 0.1 cm intervals. SD scores of body weight, height and body mass index for age Neyzi et al. It will be calculated using the reference values developed for Turkish children by Age, diabetes age, gender, height - body weight-body mass index SD score, HbA1c level, daily energy intake, percentage of energy from carbohydrate-protein-fat-saturated fat in energy, daily fiber intake amount of the cases will be recorded in the case report form. The biochemical values of the participants will be taken from the file records. The data will be entered into the statistical package program and the patients' 1) carbohydrate, protein, fat, saturated fat intake, 2) vitamin-mineral intake, and 3) fruit and vegetable consumption will be compared with the recommendations in national and international guidelines and their relationship with metabolic control will be investigated

DETAILED DESCRIPTION:
In this cross-sectional study, 150 children and adolescents with type 1 diabetes who came to Ege University Child Health and Diseases Department, Pediatric Endocrine and Diabetes Department for regular check-ups (4 diabetes control/year) and kept food consumption records in the last 1 year will be included. Body weight and height measurements of the cases will be done by the same person in Ege University Pediatric Endocrinology and Diabetes BD Polyclinic. Turkish Standard Institute approved Baster brand weighing instrument with 0.1 kg intervals and height measurements will be made with Harpander brand stadiometer with 0.1 cm intervals. SD scores of body weight, height and body mass index for age Neyzi et al. It will be calculated using the reference values developed for Turkish children by Age, diabetes age, gender, height - body weight-body mass index SD score, HbA1c level, daily energy intake, percentage of energy from carbohydrate-protein-fat-saturated fat in energy, daily fiber intake amount of the cases will be recorded in the case report form. The biochemical values of the participants will be taken from the file records. The data will be entered into the statistical package program and the patients' 1) carbohydrate, protein, fat, saturated fat intake, 2) vitamin-mineral intake, and 3) fruit and vegetable consumption will be compared with the recommendations in national and international guidelines and their relationship with metabolic control will be investigated

ELIGIBILITY:
Inclusion Criteria:

* who came to regular check-ups in the last 1 year (4 diabetes checks/year)
* children and adolescents who keep a food diary for 3 days before coming to diabetes control by their own/caregiver

Exclusion Criteria:

* Cases that do not accept to fill in the 'Informed Consent Form'
* Cases with diseases accompanying T1DM (autoimmune diseases such as celiac, cystic fibrosis, etc.)

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diabetes treatment, cases followed in Ege University Pediatrics Department, Pediatric Endocrine and Diabetes Department
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Macronutrient distribution | day 1
  The macronutrient distribution of participant's diets will be evaluated for compliance with national and international guidelines.
HbA1c | day 1
  As metabolic control parameter
Height (m), | day 1
  As a growth monitoring parameter
Weight (kg) | Day 1
  As a growth monitoring parameter
Body mass index (kg/m2) | Day 1
  As a growth monitoring parameter

CONTACTS AND LOCATIONS:
Overall Officials: yelda mansuroglu, MSc, Study Chair — Ege University; gunay demir, MSc, Study Chair — Ege University; samim ozen, Assoc Prof, Study Chair — Ege University; sukran darcan, Prof Dr, Study Chair — Ege University; damla goksen, Prof Dr, Study Director — Ege University
Locations (2):
- Turkey (Türkiye) (2):
  - Ege University, Izmir, Bornova
  - Ege University Faculty of Medicine Department of Pediatrics, Izmir

IPD SHARING:
Plan to Share IPD: Undecided